CLINICAL TRIAL: NCT02516020
Title: Effectiveness of Single Step Culture Media and Sequential Culture Media on Blastulation Rate: a Randomized Controlled Trial.
Brief Title: Effectiveness of Single Step Culture Media and Sequential Culture Media on Blastulation Rate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_ 05_2015
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Infertility
Keywords: IVF; ICSI; culture media; sequential
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Global (Active Comparator): EmbryoSingle step culture medium Embryos are cultured in single step culture from day 1 to day 5 Other Name: Global medium (LifeGlobal)
  Interventions: Drug: Global
- Origio (Active Comparator): Sequential media Embryos are cultured in sequential medium from Day1 to Day 3 and from Day 3 to Day 5 (Sequential Blast) Other Name: Sequential Blast (Origio)
  Interventions: Drug: Origio

INTERVENTIONS:
Drug: Global — Embryos are cultured in single step culture from day 1 to day 5
  Other Names: Global medium (LifeGlobal)
  Arms: Global
Drug: Origio — Embryos are cultured in sequential medium from Day1 to Day 3 and from Day 3 to Day 5 (Sequential Blast)
  Other Names: Sequential Blast (Origio)
  Arms: Origio

SUMMARY:
To compare the effectiveness of single step culture media and continuous uninterrupted culture media on blastulation rate

DETAILED DESCRIPTION:
Sequential culture media are designed to mimic the changing environment in the ovary ducts and the uterus in vivo. However, there are some differences between in vivo and in vitro culture conditions. Hence, single step media are created which allow the embryo itself to choose the necessary nutrients while maintaining a more stable culture environment. Previous studies suggest higher blastulation rate in the single step media than the sequential media.

This is an Randomized controlled trial (RCT) study comparing the blastulation rate of single step culture media and sequential culture media. Stimulation protocol is antagonist. Patient will be consulted on the day of ultrasound if they meet the inclusion criteria and sign the consent form. Then, the nurse will open the letter containing the type of media for that case. The media is prepared inside the lab a day before oocyte pick-up.

After oocyte pick-up, the oocyte-cumulus complex (OCC) will be cultured for 2 hours at 37°C, 6% Carbon dioxide (CO2) and 5% oxygen (O2). Meanwhile, sperm preparation will be performed using gradient technique. After 2 hours, OCC will be denuded and will be cultured for 1 hour until Intracytoplasmic Sperm Injection (ICSI). Oocytes after ICSI will be cultured in groups of 3-4 oocytes in the same conditions of 37 ° C, 6% CO2 and 5% O2. Fertilization check procedure is at 16-18 hours after ICSI. On day 3, the embryos will be evaluated in 66-68 hours after ICSI, grade 1 embryos are identified with 7-9 blastomeres and fragmentation is from 0-10%. The patients will be informed about the embryo quality. If the embryos are not decided to have day 5 transferring, patient will be consulted to transfer on day 3. Blastulation rate will not be recorded.

For the sequential culture media group, embryos will be transferred to Sequential Blast medium. For the single step culture media group, embryos will be transferred to the new culture dish with the same medium. On day 5, embryo quality assessment will be at 116±1 hours after ICSI. Blastocyst grading is based on the expansion, inner cell mass quality, and trophectoderm quality. Two good blastocyst will be transferred. After 11 days, beta-human chorionic gonadotropin (hCG) test will be required. If the beta-hCG result is positive, examination will be needed after 3 weeks and the luteal support will be given until 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Number of previous failure IVF cycles ≤2
* Using Gonadotropin-releasing hormone (GnRH) - Antagonist protocol for IVF
* Using GnRH for oocyte triggering.
* Read and sign consent form to participate in the study and have not been recruited for any other researches.

Exclusion Criteria:

* Oocyte donation cycles
* Abnormal uterine.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The blastulation rate | 116 ±1 hours after ICSI
  The blastulation rate is defined as the number of blastocysts from 2 pronuclei (2PN) zygotes

SECONDARY OUTCOMES:
Implantation rate | 11 days after embryo transfer
  Implantation rate is defined as the number of gestational sacs per number of embryos transferred.
Clinical pregnancy | 7 weeks after embryo transfer
  Clinical pregnancy is defined by the image gestational sac under ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — Research Center for Genetics and Reproductive Health
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam